CLINICAL TRIAL: NCT03452878
Title: Evaluation of the Functional Results of Bilateral Amygdalotomy for Refractory Aggressive Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Raquel Chacon Ruiz Martinez, Principal investigator, PhD, Hospital Sirio-Libanes
Other Study IDs: 2014-63
Record Dates: First submitted 2017-03-29; First posted 2018-03-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Aggression
Keywords: Amygdala, neurosurgery, aggressive behavior
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aggressive refractory patient: A pre defined group of individuals will be included in the study. This group is considered aggressive refractory patient and will be submitted to the bilateral amygdalotomy surgery.
  Interventions: Behavioral: Aggressive behavior

INTERVENTIONS:
Behavioral: Aggressive behavior — Aggressive Behavior Scale, Quality of Life (SF-36) and Agitated Behavior Scale, measurement of thyroid-stimulating hormone (TSH), T4, T3, Cortisol, Luteinizing Hormone (LH), Estradiol, Prolactin, Progesterone, testosterone, and sex hormone-binding globulin (SHBG) and Resonance Magnetic Imaging.

SUMMARY:
Aggressiveness has a high prevalence in the psychiatry population and is of major concern. Though pharmacological treatments are effective for most patients, there is a portion that doesn't respond properly and is considered medically refractory. For them, surgical procedures (i.e. stereotactic lesions) have been performed as an attempt to reintegrate patient into society. The amygdala is a main structure in the control of aggressive behavior and amygdala lesion could improve behavior without neurological or other behavioral impairment. In this study, it will evaluate the functional results of the bilateral amygdala lesion of aggressive refractory patients through neuroimaging, clinical assessment and blood hormonal levels. To better understand the neurobiology of aggression, aggressive patients that are not refractory will also be studied through neuroimaging and hormonal levels.

ELIGIBILITY:
Inclusion Criteria:

* Refractory aggression (Adler et al., 2015) defined by extreme levels of aggression after the use of Risperidone or Aripiprazole ou combination of others psychoactive drugs.

Exclusion Criteria:

* Patients with anatomical alterations that may disrupt the surgery, infections or non-controlled diseases, treatment with other experimental drugs, pregnant women or during lactation, psychological or sociological conditions that will not permit the patient to be accompanied by the medical staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory aggressive patients.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Aggression Levels | 48 months
  The level of aggression of the patients will be assessed using the overt aggression scale (OAS)

SECONDARY OUTCOMES:
Change in quality of life | 48 months
  The quality of life will be assessed using the quality of life scale (SF-36).
Follow-up hormones | 48 months
  The thyroid-stimulating hormone, T4, T3, luteinizing hormone, testosterone, progesterone, prolactin, estradiol, cortisol and sex hormone-binding will be evaluated. The data will be evaluate comparing to the normal range and also will be correlate with the overt aggression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Fernando Reis, PhD, Study Director — Hospital Sirio-Libanes

IPD SHARING:
Plan to Share IPD: No